CLINICAL TRIAL: NCT00458523
Title: Eradication of Minimal Residual Disease (MRD) in Patients With Chronic Lymphocytic Leukaemia (CLL) With Alemtuzumab: A Phase II Study
Brief Title: Alemtuzumab in Treating Patients With B-Cell Chronic Lymphocytic Leukemia in Partial Remission or Complete Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leeds Cancer Centre at St. James's University Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: LCC-CTRU-CLL207; CDR0000538115 (Registry Identifier: PDQ (Physician Data Query)); SPRI-LCC-CTRU-CLL207; ISRCTN23153249; EU-20715; EUDRACT-2006-000053-22
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2007-04

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; In Situ Hybridization, Fluorescence; Flow Cytometry

INTERVENTIONS:
Biological: alemtuzumab
Genetic: fluorescence in situ hybridization
Genetic: mutation analysis
Other: flow cytometry

SUMMARY:
RATIONALE: Monoclonal antibodies, such as alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them.

PURPOSE: This phase II trial is studying the side effects and how well alemtuzumab works in treating patients with B-cell chronic lymphocytic leukemia in partial remission or complete remission.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of achieving minimum residual disease (MRD) negativity after treatment with alemtuzumab in patients with B-cell chronic lymphocytic leukemia (B-CLL) who have low levels of MRD after conventional therapy or who relapse at an MRD level after a prior MRD-negative remission.
* Determine the safety of alemtuzumab in patients treated in the MRD-positive setting.

Secondary

* Determine the clinical response in patients treated with this drug.
* Determine the time to MRD relapse in patients treated with this drug.
* Determine the overall survival of patients treated with this drug.
* Determine the effect of this drug when administered as consolidation/maintenance therapy on CD52 expression on CLL cells.
* Determine the safety and efficacy of repeated drug dosing required to achieve sustained MRD negativity in these patients.

OUTLINE: This is a multicenter study.

* Observation: Patients with minimal residual disease (MRD)-negative status are observed every 4 weeks for 12 weeks and then every 12 weeks thereafter. If they become MRD-positive, then they are eligible for treatment.
* Treatment: Patients with MRD-positive status receive alemtuzumab subcutaneously or IV over 2 hours three times weekly for up to 12 weeks in the absence of disease progression or unacceptable toxicity. After completion of 6 weeks of study therapy, patients are evaluated for response. Patients who remain MRD-positive and are responding to study therapy receive an additional 6 weeks of treatment. Patients who remain MRD-positive and show no significant improvement in the level of leukemic cells detected in their peripheral blood or bone marrow are removed from the study. Patients achieving MRD-negative remission are removed from study therapy and monitored for disease recurrence at an MRD level. If MRD-level relapse is confirmed in these patients, they may be retreated with alemtuzumab provided their initial response to therapy lasted for at least 6 months.

Patients undergo collection of peripheral blood and bone marrow periodically during study for assessment of MRD by MRD flow cytometry, fluorescent in situ hybridization (FISH) analysis, somatic mutation analysis, and B-cell selection.

After completion of study therapy, patients are followed periodically.

PROJECTED ACCRUAL: A total of 54 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell chronic lymphocytic leukemia (B-CLL) meeting the following criterion:

  * Confirmed by characteristic immunophenotype on peripheral blood flow cytometry
* In complete or partial remission after prior therapy for B-CLL

  * No treatment failure after receiving prior alemtuzumab therapy
* Minimal residual disease (MRD) status meeting 1 of the following criteria:

  * Detectable B-CLL MRD (i.e., MRD-positive) as shown by peripheral blood or bone marrow involvement
  * Undetectable B-CLL MRD (i.e., MRD-negative remission)
* Lymph nodes < 2 cm in maximum diameter
* No persisting severe pancytopenia due to prior therapy rather than disease, as defined by the following criteria:

  * Neutrophil count < 5,000/mm^3
  * Platelet count < 50,000/mm^3
* No clinically progressive disease (i.e., peripheral blood B-cell count ≥ 5,000/mm³)
* No mantle cell lymphoma
* No CNS involvement with B-CLL

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy
* Creatinine < 2 times upper limit of normal (ULN)*
* Bilirubin < 2 times ULN*
* No known HIV positivity
* No concurrent active infection
* No history of anaphylaxis after exposure to rat or mouse-derived, complementary-determining region-grafted humanized monoclonal antibodies
* No other concurrent severe diseases or mental disorders
* No concurrent active secondary malignancy NOTE: *Unless secondary to direct infiltration of the liver by B-CLL or hemolysis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior allogeneic stem cell transplantation

  * Any other prior therapy allowed
* At least 6 months since completion of last therapy for B-CLL
* More than 6 weeks since prior investigational agents
* No other concurrent cytotoxic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2006-12; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Rate of undetectable minimal residual disease (MRD) after completion of alemtuzumab therapy
Rate of unacceptable toxicities

SECONDARY OUTCOMES:
Rate of overall response (complete or partial response)
Time to MRD relapse
Overall survival
Expression of CD52 on chronic lymphocytic leukemia cells
Rate of re-achievement of MRD negativity after completion of alemtuzumab therapy
Incidence of successful retreatment
Toxicity from repeated therapy
Length of interval between required treatments

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hillmen, MD, Study Chair — Leeds General Infirmary
Locations (2):
- United Kingdom (2):
  - Kent and Canterbury Hospital, Canterbury, England
  - Leeds General Infirmary, Leeds, England